CLINICAL TRIAL: NCT03805854
Title: Modulating Pain Using Transcranial Alternating Stimulation (tACS) in Healthy Human Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Technical University of Munich (Other)
Collaborators: German Research Foundation (Other)
Responsible Party: Principal Investigator, Markus Ploner, Heisenberg Professor of Human Pain Research, Technical University of Munich
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 01/2019
Record Dates: First submitted 2019-01-10; First posted 2019-01-16 (Actual); Last update posted 2020-06-04 (Actual); Status verified 2020-06

CONDITIONS: Experimental Pain in Healthy Human Subjects
Keywords: pain; tACS; alpha; gamma; neural oscillations; brain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: Each participant will participate in 6 experimental conditions aimed at studying the effect of different tACS protocols on pain processing: (1) 10 Hz tACS of the bilateral somatosensory cortex, (2) 10 Hz tACS of the prefrontal cortex, (3) 80 Hz tACS of the bilateral somatosensory cortex, (4) 80 Hz tACS of the prefrontal cortex, (5) sham stimulation of the bilateral somatosensory cortex, and (6) sham stimulation of the prefrontal cortex. Each condition will be administered in an individual session. Sessions will be conducted in pseudo-randomized order and separated by at least 24 hours to avoid any carry-over effects of the stimulation. During each tACS administration, pain will be induced by means of an established tonic thermal stimulation paradigm lasting for several minutes (TSA-II; Medoc, Ramat Yishai, Israel) while pain ratings and autonomic responses will be recorded (Nickel et al., 2017a; Nickel et al., 2017b).
Masking Description: Neither participants nor the conducting investigator will be informed about the administered tACS protocol (10 Hz tACS, 80 Hz tACS or sham stimulation) (= double-blind study). Blinding of participants will be achieved by using tACS intensities which should not evoke perceivable stimulation side effects like skin or visual sensations. Blinding of participants will be controlled using post-hoc questionnaires. An unblinded research assistant who does not interact with the participants will be responsible for initiating and monitoring the appropriate tACS protocol and, thus, enable the blinding of the conducting investigator.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Transcranial alternating current stimulation (tACS) (Experimental)
  Interventions: Device: 10 Hz tACS of the bilateral somatosensory cortex; Device: 10 Hz tACS of the prefrontal cortex; Device: 80 Hz tACS of the bilateral somatosensory cortex; Device: 80 Hz tACS of the prefrontal cortex; Device: Sham stimulation of the bilateral somatosensory cortex; Device: Sham stimulation of the prefrontal cortex

INTERVENTIONS:
Device: 10 Hz tACS of the bilateral somatosensory cortex — 10 Hz tACS at 1 mA will be applied over the bilateral somatosensory cortex for 10 minutes using a Neuroconn stimulator (DC-Stimulator MR; Neuroconn, Ilmenau, Germany) and 2 5*5 cm rubber electrodes placed at electrode positions CP3 and CP4 according to the international 10-20 system.
Device: 10 Hz tACS of the prefrontal cortex — 10 Hz tACS at 1 mA will be applied over the prefrontal cortex for 10 minutes using a Neuroconn stimulator (DC-Stimulator MR; Neuroconn, Ilmenau, Germany) and 2 5*5 cm rubber electrodes placed at electrode positions F3 and F4 according to the international 10-20 system.
Device: 80 Hz tACS of the bilateral somatosensory cortex — 80 Hz tACS at 1 mA will be applied over the bilateral somatosensory cortex for 10 minutes using a Neuroconn stimulator (DC-Stimulator MR; Neuroconn, Ilmenau, Germany) and 2 5*5 cm rubber electrodes placed at electrode positions CP3 and CP4 according to the international 10-20 system.
Device: 80 Hz tACS of the prefrontal cortex — 80 Hz tACS at 1 mA will be applied over the prefrontal cortex for 10 minutes using a Neuroconn stimulator (DC-Stimulator MR; Neuroconn, Ilmenau, Germany) and 2 5*5 cm rubber electrodes placed at electrode positions F3 and F4 according to the international 10-20 system.
Device: Sham stimulation of the bilateral somatosensory cortex — 10 Hz tACS at 1 mA will be applied over the bilateral somatosensory cortex for 10 seconds at the beginning of the experimental session using a Neuroconn stimulator (DC-Stimulator MR; Neuroconn, Ilmenau, Germany) and 2 5*5 cm rubber electrodes placed at electrode positions CP3 and CP4 according to the international 10-20 system.
Device: Sham stimulation of the prefrontal cortex — 10 Hz tACS at 1 mA will be applied over the prefrontal cortex for 10 seconds at the beginning of the experimental session using a Neuroconn stimulator (DC-Stimulator MR; Neuroconn, Ilmenau, Germany) and 2 5*5 cm rubber placed at electrode positions F3 and F4 according to the international 10-20 system.

SUMMARY:
Pain is a highly complex and subjective phenomenon which results from the dynamic integration of sensory and contextual (i.e. cognitive, emotional, and motivational) processes. Recent evidence suggests that neural oscillations and their synchronization between different brain areas might form the basis of these integrative functions. When investigating tonic experimental pain lasting for several minutes, for example, objective stimulus intensity is inversely related to alpha (8-13 Hz) and beta (13-30 Hz) oscillations in early somatosensory areas, while subjective pain intensity is positively associated with gamma (30-100 Hz) oscillations in prefrontal cortex. Yet, with a few exemptions, reported links between oscillatory brain activity and pain have mostly been established by correlative approaches which do not allow to infer causality. The current project aims at comprehensively investigating the causal role of neural oscillations for tonic experimental pain in healthy human subjects. To this end, transcranial alternating current stimulation (tACS) will be employed to modulate oscillatory brain activity in alpha and gamma frequency bands and investigate effects of this manipulation on pain perception and pain-related autonomic responses. Using an established tonic pain stimulation protocol and a double-blind, sham-controlled design, effects of tACS of somatosensory as well as prefrontal brain areas will be investigated. Results promise to elucidate the neural mechanisms underlying tonic experimental pain by testing the mechanistic role of neural oscillations in different aspects of pain processing. Furthermore, they might contribute to the development of urgently needed new treatment approaches for chronic pain using neuromodulatory methods.

ELIGIBILITY:
Inclusion Criteria:

* aged 18-65 years
* Right-handedness
* Written informed consent

Exclusion Criteria:

* Pregnancy
* Neurological or psychiatric diseases (e.g. epilepsy, stroke, depression, anxiety disorders)
* Severe general illnesses (e.g. tumors, diabetes)
* Skin diseases (e.g. dermatitis, psoriasis or eczema)
* Current or recurrent pain
* Regular intake of medication
* Surgical procedures involving the head or spinal cord
* Head trauma followed by impairment of consciousness
* Past fainting spells or syncopes
* Metal (except titanium) or electronic implants
* Side-effects following previous electrical or magnetic stimulation
* Side-effects following previous thermal stimulation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2019-04-15 (Actual); Primary Completion 2019-10-23 (Actual); Study Completion 2019-10-23 (Actual)

PRIMARY OUTCOMES:
Changes in pain rating on visual analogue scale (VAS; 0: 'no pain' to 10: 'maximal tolerable pain') between sessions | During 10 min thermal stimulation in each of six interventions (10 Hz tACS/80 Hz tACS/sham stimulation of the somatosensory/prefrontal cortex), which are separated by at least 24 hrs.
  During thermal stimulation, participants will be instructed to continuously rate the currently perceived pain intensity using a finger-span device.
Changes in skin conductance responses (µS) between sessions | During 10 min thermal stimulation in each of six interventions (10 Hz tACS/80 Hz tACS/sham stimulation of the somatosensory/prefrontal cortex), which are separated by at least 24 hrs.
  Skin conductance responses will be recorded using two electrodes attached to the index and middle finger of the left hand.
Changes in heart rate (BPM, beats per minute) between sessions | During 10 min thermal stimulation in each of six interventions (10 Hz tACS/80 Hz tACS/sham stimulation of the somatosensory/prefrontal cortex), which are separated by at least 24 hrs.
  The electrocardiogram (ECG) will be recorded using two electrodes placed under the right clavicle and below the sternum, respectively.
Changes in oscillatory brain activity before and after tACS application within each session | Measured immediately before and after the tACS protocol in each of six interventions (10 Hz tACS/80 Hz tACS/sham stimulation of the somatosensory/prefrontal cortex), which are separated by at least 24 hrs.
  5-minute resting state electroencephalogram (EEG) will be recorded with two electrodes placed at the same electrode positions used for the respective tACS protocol. Power of oscillatory brain activity will be quantified in the alpha (8-12 Hz) and gamma (30-100 Hz) bands.

SECONDARY OUTCOMES:
Perception of tACS induced visual and skin sensations measured by numerical rating scale (NRS; 0: 'no sensation' to 10: 'very strong sensation') | Measured immediately after the EEG measurement following each of six interventions (10 Hz tACS/80 Hz tACS/sham stimulation of the somatosensory/prefrontal cortex), which are separated by at least 24 hrs.
  The perception of visual and skin sensations induced by the tACS protocols will be assessed using a custom questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Markus Ploner, Prof. Dr. med., Principal Investigator — Department of Neurology, Klinikum rechts der Isar, Technische Universität München
Locations (1):
- Department of Neurology, Klinikum rechts der Isar, Technische Universität München, Munich, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: Yes
Pseudonymized individual participant data sets will be made available at the OSF online repository [https://osf.io/] upon publication.
URL: https://osf.io/pnd6g/

REFERENCES:
- [Background] Ahn S, Prim JH, Alexander ML, McCulloch KL, Frohlich F. Identifying and Engaging Neuronal Oscillations by Transcranial Alternating Current Stimulation in Patients With Chronic Low Back Pain: A Randomized, Crossover, Double-Blind, Sham-Controlled Pilot Study. J Pain. 2019 Mar;20(3):277.e1-277.e11. doi: 10.1016/j.jpain.2018.09.004. Epub 2018 Sep 27. PMID 30268803
- [Background] Arendsen LJ, Hugh-Jones S, Lloyd DM. Transcranial Alternating Current Stimulation at Alpha Frequency Reduces Pain When the Intensity of Pain is Uncertain. J Pain. 2018 Jul;19(7):807-818. doi: 10.1016/j.jpain.2018.02.014. Epub 2018 Mar 15. PMID 29551661
- [Background] Herrmann CS, Rach S, Neuling T, Struber D. Transcranial alternating current stimulation: a review of the underlying mechanisms and modulation of cognitive processes. Front Hum Neurosci. 2013 Jun 14;7:279. doi: 10.3389/fnhum.2013.00279. eCollection 2013. PMID 23785325
- [Background] Jensen MP, Day MA, Miro J. Neuromodulatory treatments for chronic pain: efficacy and mechanisms. Nat Rev Neurol. 2014 Mar;10(3):167-78. doi: 10.1038/nrneurol.2014.12. Epub 2014 Feb 18. PMID 24535464
- [Background] Nickel MM, May ES, Tiemann L, Postorino M, Ta Dinh S, Ploner M. Autonomic responses to tonic pain are more closely related to stimulus intensity than to pain intensity. Pain. 2017 Nov;158(11):2129-2136. doi: 10.1097/j.pain.0000000000001010. PMID 28700538
- [Background] Nickel MM, May ES, Tiemann L, Schmidt P, Postorino M, Ta Dinh S, Gross J, Ploner M. Brain oscillations differentially encode noxious stimulus intensity and pain intensity. Neuroimage. 2017 Mar 1;148:141-147. doi: 10.1016/j.neuroimage.2017.01.011. Epub 2017 Jan 7. PMID 28069543
- [Background] Ploner M, Sorg C, Gross J. Brain Rhythms of Pain. Trends Cogn Sci. 2017 Feb;21(2):100-110. doi: 10.1016/j.tics.2016.12.001. Epub 2016 Dec 23. PMID 28025007
- [Background] Polania R, Nitsche MA, Ruff CC. Studying and modifying brain function with non-invasive brain stimulation. Nat Neurosci. 2018 Feb;21(2):174-187. doi: 10.1038/s41593-017-0054-4. Epub 2018 Jan 8. PMID 29311747
- [Background] Schulz E, May ES, Postorino M, Tiemann L, Nickel MM, Witkovsky V, Schmidt P, Gross J, Ploner M. Prefrontal Gamma Oscillations Encode Tonic Pain in Humans. Cereb Cortex. 2015 Nov;25(11):4407-14. doi: 10.1093/cercor/bhv043. Epub 2015 Mar 8. PMID 25754338
- [Background] Sitaram R, Ros T, Stoeckel L, Haller S, Scharnowski F, Lewis-Peacock J, Weiskopf N, Blefari ML, Rana M, Oblak E, Birbaumer N, Sulzer J. Closed-loop brain training: the science of neurofeedback. Nat Rev Neurosci. 2017 Feb;18(2):86-100. doi: 10.1038/nrn.2016.164. Epub 2016 Dec 22. PMID 28003656
- [Background] Vosskuhl J, Struber D, Herrmann CS. Non-invasive Brain Stimulation: A Paradigm Shift in Understanding Brain Oscillations. Front Hum Neurosci. 2018 May 25;12:211. doi: 10.3389/fnhum.2018.00211. eCollection 2018. PMID 29887799
- [Derived] May ES, Hohn VD, Nickel MM, Tiemann L, Gil Avila C, Heitmann H, Sauseng P, Ploner M. Modulating Brain Rhythms of Pain Using Transcranial Alternating Current Stimulation (tACS) - A Sham-Controlled Study in Healthy Human Participants. J Pain. 2021 Oct;22(10):1256-1272. doi: 10.1016/j.jpain.2021.03.150. Epub 2021 Jun 12. PMID 33845173